CLINICAL TRIAL: NCT06872606
Title: The Efficacy and Safety of Short-Course Radiotherapy Combined with Intracavitary Brachytherapy Followed by Pucotenlimab, Bevacizumab, Oxaliplatin, and Trifluridine/Tipiracil (TAS-102) for Total Neoadjuvant Therapy of Microsatellite Stable (MSS) Locally Advanced Low Rectal Adenocarcinoma: an Prospective, Single Arm Clinical Trial （SCRIPBOT Trial）
Brief Title: Short-Course Radiotherapy Combined with Intracavitary Brachytherapy Followed by Pucotenlimab, Bevacizumab, Oxaliplatin, and Trifluridine/Tipiracil (TAS-102) for Total Neoadjuvant Therapy of Microsatellite Stable (MSS) Locally Advanced Low Rectal Cancer
Acronym: SCRIPBOT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Sheng Dai, Director, Medical affairs department, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0623
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Rectal Adenocarcinoma
Keywords: Short-Course Radiotherapy; Pucotenlimab; Oxaliplatin; Bevacizumab; Trifluridine/Tipiracil（TAS-102）
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Trifluridine; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- POBTAS Trial Arm (Experimental): Intervention:
  1.Radiotherapy:
  1. Phase 1 (Short-Course External Radiotherapy):
     Intensity-modulated radiotherapy (IMRT) at 5 Gy X 5F, completed within 1 week.
  2. Phase 2 (Intracavitary Brachytherapy):
  Administered during weeks 5-6, targeting residual lesions with 3Gy X 3F, completed within 1 week.
  2.Systemic Therapy Post-Initial Radiotherapy:
  1. Cycles 1-2: PD-1 antibody immunotherapy (pucotenlimab) combined with bevacizumab, oxaliplatin, and trifluridine/tipiracil (TAS-102).
  2. Cycles 3-4: Sequential PD-1 immunotherapy + oxaliplatin + TAS-102 (bevacizumab omitted in Cycle 4).
  3.Post-Cycle 4 Evaluation: If ypT0 (local pathological complete response): Enter follow-up observation. If non-CR: Proceed to Step 4.
  4.Extended Systemic Therapy for Non-CR Patients: Cycles 5-8: Repeat PD-1 immunotherapy + bevacizumab + oxaliplatin + TAS-102 (bevacizumab omitted in Cycle 8).
  5.Post-Cycle 8 Evaluation: If ypT0: Enter follow-up observation. If non-ypT0: Proceed to TME surgery.
  Interventions: Drug: Pucotenlimab; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Trifluridine/Tipiracil Hydrochloride; Radiation: Short-course radiotherapy; Radiation: intracavitary brachytherapy

INTERVENTIONS:
Drug: Pucotenlimab — Pucotenlimab (200 mg IV, q3w)
Drug: Bevacizumab — Bevacizumab (7.5 mg/kg IV, q3w)
Drug: Oxaliplatin — Oxaliplatin (130 mg/m² IV, q3w)
Drug: Trifluridine/Tipiracil Hydrochloride — TAS-102 (25 mg/m² orally, days 1-5 and 8-12).
Radiation: Short-course radiotherapy — (25 Gy/5 fractions)
Radiation: intracavitary brachytherapy — brachytherapy (3 Gy/3 fractions).

SUMMARY:
A Prospective Single-Arm Study of Short-Course Radiotherapy Followed by PD-1 Monoclonal Antibody, Bevacizumab, Oxaliplatin, and Trifluridine/Tipiracil for Total Neoadjuvant Therapy in MSS Locally Advanced Low Rectal Cancer. This is a Non-Randomized, Single Group Assignment, Open Label, Phase: Phase II study. The Primary Objective is to assess the organ preservation rate (clinical complete response, cCR) after total neoadjuvant therapy. Secondary Objectives are Tumor regression grade (TRG), 3-year overall survival (OS) and disease-free survival (DFS), and Safety and quality of life (QoL). In this study, the investigators will perform the multi-dimensional omics study to explore the tumors microenvironments, explore the characteristics of the treatment benefit population, and try to construct an efficacy prediction model to screen the treatment benefit population early and implement precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to receive neoadjuvant therapy.
2. ≧18 years old.
3. Diagnosed by digital rectal examination, colonoscopy, and high-resolution MRI of the pelvis, the tumor is less than or equal to 5 cm from the anus.
4. Histologically diagnosed as rectal adenocarcinoma.
5. Clinical stage: cT2-4a N+ or cT3/T4a N0 (MRI/CT-confirmed).
6. MSS/pMMR status confirmed by immunohistochemistry or PCR before treatment .
7. ECOG Scale of Performance Status score 0-1 point.
8. Adequate organ function (hematologic, hepatic, renal).
9. Have not received anti-tumor and immunotherapy before enrollment.
10. Laboratory inspections must meet the following standards:

1) White blood cell count>3.5×109/L, absolute value of neutrophils>1.8×109/L, platelet count ≥75×109/L, hemoglobin ≥100g/L; 2) INR≤1.5, and APTT≤1.5 times the upper limit of normal or partial prothrombin time (PT) ≤1.5 times the upper limit of normal; 3) Total bilirubin ≤ 1.25 times the upper limit of normal; ALT and AST < 5 times the upper limit of normal; 4) 24h creatinine clearance >50mL/min or serum creatinine <1.5 times the upper limit of normal.

11. Voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. History of other malignant diseases in the past 5 years.
2. Patients with metastases from other sites (stage IV patients).
3. Patients withT4b or positive lateral lymph nodes by pelvic contrast-enhanced CT and pelvic high-resolution MRI.
4. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. requiring emergency surgery.
5. Known allergic to oxaliplatin, PD-1 monoclonal antibody and other intervention drugs.
6. Pathologically suggested signet ring cell carcinoma and mucinous adenocarcinoma.
7. dMMR or MSI-H patients.
8. The patient is accompanied by any unstable systemic disease, including but not limited to: severe infection, uncontrolled diabetes, hypertension uncontrolled by medication, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardial Infarction, congestive heart failure, severe cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease; disease affecting the patient's life.
9. The disease (such as mental illness, etc.) or condition (such as alcoholism or drug abuse, etc.) associated with the patient will increase the risk of the patient receiving the trial drug treatment or affect the patient's compliance with the trial requirements, or may confuse the research results.
10. Active autoimmune disease that may worsen while receiving immunostimulants.
11. Known history of positive HIV test or known acquired immunodeficiency syndrome.
12. Patients who are using immunosuppressive agents, except for the following conditions:

1) Intranasal, inhaled, topical steroids, or topical steroid injections (eg, intra-articular injections); 2) Physiological doses of systemic corticosteroids ≤10 mg/day prednisone or equivalent; 3) Steroids used to prevent allergic reactions (eg, before CT scan). 13. Received any other experimental drug treatment or participated in another interventional clinical trial within 30 days before screening 14. Women who are pregnant or breastfeeding or who plan to become pregnant or breastfeeding during the study period; men or women who are unwilling to take effective contraceptive measures.

15. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, etc.

16. Other conditions that the investigator judges that the patient is not suitable to participate in the clinical study, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Organ preservation rate | Up to 2 weeks (once evaluation or biopsy is done)
  The organ preservation rate was calculated as the percentage of participants who achieved cCR and were spared from total mesorectal excision (TME) surgery relative to the total study cohort. Clinical complete response (cCR) requires both histopathological confirmation (no viable tumor cells in biopsy specimens) and radiographic confirmation (absence of tumor on CT, MRI, or PET-CT).

SECONDARY OUTCOMES:
Total mesorectal excision rate | After 2 weeks (once biopsy or local excision is done)
  Population who not achieve complete clinical response and have TME surgery after total neoadjuvant therapy
Total mesorectal excision rate after recurrence | Through study completion, an average of 3 year
  Population who recurrent and have Salvage total mesorectal excision after achieving complete clinical response after total neoadjuvant therapy
Tumor regression grade | After 2 weeks (once biopsy or local excision is done)
  Tumor Regression Grade（TRG）will be done via pathologic assessment on the surgical specimen with AJCC/CAP TRG system
Overall survival | Up to 3 years
  The proportion of participants who remain survival at 3 years
Progression free survival | Up to 3 years
  The proportion of participants who remain progression free at 3 years
TRAEs | Up to 3 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0
Surgical Complications | Up to 3 years
  Surgical Complications of biopsy, local excision or total mesorectal resection procedure for patients as assessed by Clavien-Dindo classification.
QoL | Up to 3 years
  Quality of life of the patients in total neoadjuvant settings as assessed by Functional Assessment of Cancer Therapy - Colorectal (FACT-C) questionnaire liscenced from The Functional Assessment of Chronic Illness Therapy System ("FACIT System"). By using the Manual scoring template, some items are reverse scored. Subscale scores, total scores and TOI scores. The higher the score, the better the QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided